CLINICAL TRIAL: NCT06656013
Title: The Effect of Motivational Interviewing on the Level of Nomophobia and Smartphone Addiction of Nursing Students
Brief Title: Motivational Interview and Nomophobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Ayaz Alkaya (Other)
Responsible Party: Sponsor-Investigator, Sultan Ayaz Alkaya, Prof. Dr., Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024 - 954
Record Dates: First submitted 2024-10-09; First posted 2024-10-24 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Nomophobia; Smartphone Addiction
Keywords: nursing student; smartphone addiction; nomophobia; motivational interview
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interview (Experimental): Preparation and motivational interviewing practice consisting of 4 sessions
  Interventions: Behavioral: Motivational Interview
- Control (No Intervention): There will be no intervention

INTERVENTIONS:
Behavioral: Motivational Interview — After the preparation session, 4 sessions of motivational interviewing will be applied. Motivational interviewing techniques will be used in the interviews to target behavioral change.
  Arms: Motivational Interview

SUMMARY:
A preparation session and a motivational interview consisting of 4 sessions will be applied to nursing students. Data collection tools will be applied before, after and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years of age
* being a first-year nursing student
* agreeing to participate in the research

Exclusion Criteria:

* having problems understanding and speaking Turkish
* having visual or hearing impairment
* having a neuropsychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Nomophobia Scale | Pre-test
  The scale, developed by Yıldırım and Correira (2015) and adapted to Turkish by Yıldırım et al. (2016), is itemized according to the 7-point Likert type. The scale consists of 20 items and is graded as 1 = strongly disagree, 7 = strongly agree. The total score of the scale is between 20-140. A score range of 0-20 indicates that the individual does not have nomophobia, a score range of 21-60 indicates that the individual has a low level of nomophobia, a score range of 61-100 indicates that the individual has a moderate level of nomophobia, and a score range of 101-140 indicates that the individual has a high level of nomophobia.
Smartphone Addiction Scale-Short Form | Pre-test
  The Turkish validity and reliability study was conducted by Noyan et al. (2015). The scale consisting of 10 questions is evaluated with a 6-point Likert scale. Scale items are graded as "(1) Strongly disagree, (2) Disagree, (3) Partially disagree, (4) Partially agree, (5) Agree, (6) Strongly agree." The total score of the scale varies between 10 and 60, and scores above 32 indicate smartphone addiction.
Nomophobia Scale | 6 weeks after pre-test
  The scale, developed by Yıldırım and Correira (2015) and adapted to Turkish by Yıldırım et al. (2016), is itemized according to the 7-point Likert type. The scale consists of 20 items and is graded as 1 = strongly disagree, 7 = strongly agree. The total score of the scale is between 20-140. A score range of 0-20 indicates that the individual does not have nomophobia, a score range of 21-60 indicates that the individual has a low level of nomophobia, a score range of 61-100 indicates that the individual has a moderate level of nomophobia, and a score range of 101-140 indicates that the individual has a high level of nomophobia.
Smartphone Addiction Scale-Short Form | 6 weeks after pre-test
  The Turkish validity and reliability study was conducted by Noyan et al. (2015). The scale consisting of 10 questions is evaluated with a 6-point Likert scale. Scale items are graded as "(1) Strongly disagree, (2) Disagree, (3) Partially disagree, (4) Partially agree, (5) Agree, (6) Strongly agree." The total score of the scale varies between 10 and 60, and scores above 32 indicate smartphone addiction.
Nomophobia Scale | Follow-up (18 weeks after pre-test)
  The scale, developed by Yıldırım and Correira (2015) and adapted to Turkish by Yıldırım et al. (2016), is itemized according to the 7-point Likert type. The scale consists of 20 items and is graded as 1 = strongly disagree, 7 = strongly agree. The total score of the scale is between 20-140. A score range of 0-20 indicates that the individual does not have nomophobia, a score range of 21-60 indicates that the individual has a low level of nomophobia, a score range of 61-100 indicates that the individual has a moderate level of nomophobia, and a score range of 101-140 indicates that the individual has a high level of nomophobia.
Smartphone Addiction Scale-Short Form | Follow-up (18 weeks after pre-test)
  The Turkish validity and reliability study was conducted by Noyan et al. (2015). The scale consisting of 10 questions is evaluated with a 6-point Likert scale. Scale items are graded as "(1) Strongly disagree, (2) Disagree, (3) Partially disagree, (4) Partially agree, (5) Agree, (6) Strongly agree." The total score of the scale varies between 10 and 60, and scores above 32 indicate smartphone addiction.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No